CLINICAL TRIAL: NCT06057259
Title: Comparison of the Validity and Reliability of Three Different Methods Used for Wrist Proprioception Measurement
Brief Title: Validity and Reliability of Wrist Proprioception Measurement Methods
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Barış SEVEN, Ph.D. research assistant, Gazi University
Other Study IDs: 3
Record Dates: First submitted 2023-09-06; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Position Sense Disorders; Wrist
Keywords: joint; hand; sensation; Therapy; Occupational
MeSH Terms: conditions — Somatosensory Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Inclinometer: Measuring Wrist Joint Position Sense with a Inclinometer
  Interventions: Device: Joint position sense measurement
- Goniometer: Measuring Wrist Joint Position Sense with a Goniometer
  Interventions: Device: Joint position sense measurement
- Joint position sense goniometer: Measuring Wrist Joint Position Sense with a joint position sense goniometer
  Interventions: Device: Joint position sense measurement

INTERVENTIONS:
Device: Joint position sense measurement — The participants' wrist joint position sense was evaluated.

SUMMARY:
The goal of this observational study is to compare the validity and reliability of three Different methods used for wrist proprioception measurement in the healthy population. The main question[s] it aims to answer are:

* Are the methods valid and reliable?
* Which method is superior?

Wrist proprioception measurement of the participants is performed. Researchers compared the inclinometer, goniometer, and joint position sense goniometer to determine the superior method.

DETAILED DESCRIPTION:
Proprioception is one of the most important mechanisms involved in ensuring the optimal position of the wrist to prevent injuries. It occurs through stimuli from different structures such as muscle, tendon, joint capsule and skin and provides the perception of the joint's position and movement characteristics (direction, speed, etc.). This perception is essential for effective and safe motor performance. Previous studies have provided evidence that proprioceptive training yields improvements in somatosensory and sensorimotor function. Furthermore, a relationship between the loss of proprioception and motor function has also been demonstrated. Additionally, proprioceptive training reduces the frequency of injuries and provides a faster and more efficient rehabilitation process. Therefore, it is essential to detect proprioceptive defects as a part of patient evaluation which is only achievable by using valid and reliable assessment tools.

Proprioception encompasses both static (i.e., joint position sense (JPS)) and dynamic (i.e., kinesthesia) components of joint perception. Many tools and methods are available to evaluate these components, including universal goniometer, inclinometer, wrist goniometer, mobile applications, robot-assisted assessment, and isokinetic dynamometers. Especially, goniometer, inclinometer, and isokinetic dynamometer are widely used in evaluating proprioception. However, the number of studies on the validity and reliability of these tools is very limited for the wrist. In addition to these tools, the joint position sense goniometer (JPSG) is replicated and used by researchers due to its low cost and accessibility.

Although some studies found goniometer to have high precision in wrist trauma patients, there are still no gold standard tests or tools available for evaluating wrist proprioception. Therefore, it becomes confusing for researchers and clinicians to decide which method should be used in their practice accurately. In line with all these data, the present study aimed to examine the validity and test-retest reliability of two frequently used methods (Goniometer and Inclinometer) and JPSG in wrist proprioception assessment.

The detailed information about the measurements is provided in the "Study Protocol" file.

ELIGIBILITY:
Inclusion Criteria:

* After providing detailed information about the study, individuals who had agreed to participate in the research were included in the study

Exclusion Criteria:

* individuals who suffered an injury or underwent a surgical procedure in the last six months that could affect hand functions or senses were excluded from the study.
* Individuals with a history of neuromuscular disease, traumatic nerve injury, congenital anomalies, or skin infections were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteer participants
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2019-04-12 (Actual); Study Completion 2019-06-09 (Actual)

PRIMARY OUTCOMES:
Active joint position sense measurement with the Goniometer | through study completion, an average of 1 year
  The goniometric (1° scale increments) measurement was performed with the elbow positioned at 90° flexion and resting on the table, the forearm was in mid-pronation, and the fingers were relaxed. The movement axis of the mid-carpal and radiocarpal joints is defined as the pivot point of the goniometer to ensure a compatible measurement of wrist movement. The stable arm of the goniometer was placed parallel to the radius, and the mobile arm followed the third metacarpal bone.
Active joint position sense measurement with the Joint Position Sense Goniometer | through study completion, an average of 1 year
  The JPSG consists of two wooden boards fixed at an angle of 90°. The plate perpendicular to the ground has an opening that the wrist can go through. 0 to 180° angle values with 1° increments were drawn on the plate that parallels the floor. For the evaluation, the participant was asked to sit in front of the table with the trunk upright and the shoulder in the neutral position. The patient's forearm passed through the opening in the JPSG, and the wrist joint was adjusted to match the axis of movement. The forearm was positioned in mid-pronation, the wrist was positioned at 0° flexion/extension, and the forearm was in the neutral position. Participants were asked not to contact the plates during the measurements.
Active joint position sense measurement with the Inclinometer | through study completion, an average of 1 year
  Another tool used to evaluate wrist active joint position sense was the digital dual inclinometer. The limb position used during the inclinometer evaluations was the same as the position for the goniometer. One of the inclinometer sensors was placed on the 3rd metacarpal bone on the dorsal side of the hand. The other sensor was placed on the dorsal side of the forearm, perpendicular to the flexion/extension movement axis.

SECONDARY OUTCOMES:
Active joint position sense measurement with the Cybex Isokinetic Dynamometer | through study completion, an average of 1 year
  The Cybex isokinetic dynamometer was used as a reference standard to test the validity of the methods. The evaluation of proprioception using the isokinetic dynamometer was performed with the participants in sitting. The shoulder was positioned in the midline, the elbow was flexed about 90°, and the wrist was positioned in supination. During the evaluation, the forearm was fixed with a strap to prevent the forearm from moving and changing the angle of the wrist. The rotation axis of the dynamometer was aligned with the diagonal axis of the distal tubercule of radius and the head of ulna. The wrist was placed in a 0° position. In this starting position, the range of motion was set as 40° flexion and 40°extension. The device was calibrated before the evaluation of each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Barış SEVEN, Ph.D, Principal Investigator — İzmir Katip Çelebi University
Locations (1):
- Barış SEVEN, Izmir, Çiğli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2018-06-25): https://cdn.clinicaltrials.gov/large-docs/59/NCT06057259/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-25): https://cdn.clinicaltrials.gov/large-docs/59/NCT06057259/SAP_001.pdf